CLINICAL TRIAL: NCT04575025
Title: Special Drug Use-results Surveillance of Tabrecta Tablets (MET Exon 14 Skipping Mutation-positive Unresectable Advanced/Recurrent Non-small Cell Lung Cancer)
Brief Title: Special Drug Use-results Surveillance of Tabrecta Tablets
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280AJP01
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; non-small cell lung cancer; MET exon 14 skipping mutation-positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tabrecta tablets: Patients administered Tabrecta by prescription
  Interventions: Drug: Tabrecta tablets

INTERVENTIONS:
Drug: Tabrecta tablets — There was no treatment allocation. Patients administered Tabrecta by prescription that had started before inclusion of the patient into the study were enrolled.

SUMMARY:
This study was an uncontrolled, primary data collection-based observational study to be conducted as a central registration system, multicenter special drug-use results surveillance. As an all-case study, this study collected all patients treated with Tabrecta in a specified post-marketing period. The observation period of each patient was up to 1 year (52 weeks)

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving Tabrecta for MET exon 14 skipping mutation-positive unresectable advanced/recurrent NSCLC during a specified post-marketing period

Exclusion Criteria:

-

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving Tabrecta for MET exon 14 skipping mutation-positive unresectable advanced/recurrent NSCLC during a specified post-marketing period. By allowing patients who started Tabrecta administration before the conclusion of a contract for this study to be included in the study population after the contract, all patients treated with Tabrecta were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse reactions | 1 year
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Tabrecta or whose causality is not recorded.
Response rate | 1 year
  A response rate is defined as a proportion of patients whose best overall response is CR or PR as assessed by the RECIST version 1.1(Eisenhauer et al. 2009). Patients assessed as not evaluable (NE) were handled as non-responders, and included in the denominator for the calculation of response rates.
Overall survival rate | 1 year
  The Kaplan-Meier method was used to estimate the survival curve. Overall survival is defined as the duration from the start date of Tabrecta administration to death of any cause. For patients surviving to the end, OS was censored at the end date of the observation period.
Progression-free survival (PFS) | 1 year
  the Kaplan-Meier method was used to estimate the PFS curve according to RECIST version 1.1 (Eisenhauer et al. 2009).
  PFS is defined as the duration from the start date of Tabrecta administration to the date of the date of the first PD observed or death of any cause, whichever comes first. For patients without these events, PFS was censored at the end date of the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (63):
- Japan (63):
  - Novartis Investigative Site, Kōnan, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Okazaki, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Daisen, Akita
  - Novartis Investigative Site, Hachinohe, Aomori
  - Novartis Investigative Site, Sakura, Chiba
  - Novartis Investigative Site, Fukui-shi, Fukui
  - Novartis Investigative Site, Yoshida-gun, Fukui
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Higashihiroshima, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kan’onjichō, Kagawa-ken
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Kumagaya, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Edogawa City, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Minato, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Tama, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Higashi Okitama, Yamagata
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18351